CLINICAL TRIAL: NCT03238560
Title: Population Pharmacokinetics of Montelukast in Infants and Children
Brief Title: The Population Pharmacokinetics of Montelukast in Infants and Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Other Study IDs: 2016Montelukast001
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Montelukast Chewable Tablet — Montelukast treatment was used at a dosage of 5mg/day once daily

SUMMARY:
The investigators' aim was to evaluate the population pharmacokinetics of montelukast in infants and children and define the appropriate dose in order to optimize Montelukast treatment in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* patients have been diagnosed with asthma; age range: 1 month to 12 years old; montelukast used as part of regular treatment.

Exclusion Criteria:

* expected survival time less than the treatment cycle; patients with other factors that researcher considers unsuitable for inclusion.

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The patients are cared in the department of pediatric respiratory at Shandong Provincial Qianfoshan Hospital, Jinan, China.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
plasma concentration | 3(2-4) h, 8(6-10) h, 22 (20-24) h after oral administration
  To detect the plasma concentrations of montelukast at 3(2-4) h, 8(6-10) h, 22 (20-24) h after oral administration.
bronchoalveolar lavage fluid(BALF) | Procedure (When the patient underwent fiberoptic bronchoscopy)
  To detect the concentrations of montelukast in bronchoalveolar lavage fluid

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Ph.D, Principal Investigator — Shandong University
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Ji'nan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided